CLINICAL TRIAL: NCT02873572
Title: Marqueurs de vulnérabilité Aux Jeux Pathologiques
Brief Title: Vulnerability Markers in Pathological Gambling
Acronym: GambleMMORe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Saint Anne's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: N/2009/54
Record Dates: First submitted 2016-08-12; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Gaming; Gambling
Keywords: Online poker; Casino; Massively Multiplayer Online Role-Playing Game (MMORPG); Iowa Gambling Task (IGT); High Resolution Electroencephalography (HR-EEG)
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- online poker gamblers (Experimental): Recruitment by forums of online poker gamblers: an explanation of the research is sent with the dedicated link of the research.
  Interventions: Behavioral: step 1: online assessment; Behavioral: step2: biomarkers of gamblers/gamers
- casino gamblers (Experimental): Recruitment to the casino gates: an explanation of the research is sent with the dedicated e-link of the research and they could answer directly to the questionnaire (1st step) on sites.
  Interventions: Behavioral: step 1: online assessment; Behavioral: step2: biomarkers of gamblers/gamers
- MMORPG gamers (Experimental): Recruitment by forums of MMORPG (as guilds): an explanation of the research is sent with the dedicated link of the research.
  Interventions: Behavioral: step 1: online assessment; Behavioral: step2: biomarkers of gamblers/gamers
- no gamer subjects (Experimental): Recruitment by poster.
  Interventions: Behavioral: step 1: online assessment; Behavioral: step2: biomarkers of gamblers/gamers

INTERVENTIONS:
Behavioral: step 1: online assessment — Anonymous psychiatric and behavioral assessments to evaluate in particular addiction or pathological gambling/gaming and behavioral profile of gamblers/gamers. Once questionnaire completed, if the subjects want to continue to participate, they sent their email to investigators.
Behavioral: step2: biomarkers of gamblers/gamers — For each arm, subjects were divided into 2 groups: dependant or not dependant gamblers/gamers. Investigators focused on decision-making biomarkers following the following flow-chart:
  * psychiatric assesment and
  * registration of brain activity during a decision-making task in conditions of uncertainty (IGT) with its version for HR-EEG validated by investigators (Giustiniani, 2015).

SUMMARY:
Addictions without substances are an emergent problem giving rise to a recent and increasing request of care. Among these new addictions, pathological gambling and pathological online video gaming which are up. The purpose of this study is to identify vulnerability factors (personality traits, decision making strategies...), which are common or specific to each type of game (on line poker, casino, MMORPG, and no-gamers).

ELIGIBILITY:
Inclusion Criteria:

* arm 1: online poker gamblers who don't play another type of gamble/game
* arm 2: casino gamblers who don't play another type of gamble/game
* arm 3: MMORPG gamers who don't play another type of gamble/game
* arm 4: no-gamblers/gamers subjects
* step 2 : only right-handled subjects (due to registration of brain activity)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-04; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Compare the average activation differences in each arm regarding the dependance level and between the 4 arms. | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gorwood, MD PhD, Principal Investigator — Saint Anne's Hospital
Locations (1):
- CHU Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giustiniani J, Gabriel D, Nicolier M, Monnin J, Haffen E. Neural Correlates of Successful and Unsuccessful Strategical Mechanisms Involved in Uncertain Decision-Making. PLoS One. 2015 Jun 18;10(6):e0130871. doi: 10.1371/journal.pone.0130871. eCollection 2015. PMID 26086196